CLINICAL TRIAL: NCT02991846
Title: A Prospective Observational Study for Evaluating Incidence, Severity and Outcomes of Chronic Graft-versus-Host Disease According to 2015 NIH Consensus Criteria
Brief Title: A Prospective Observational Study for Evaluating CGVHD
Acronym: GITMO-GVCrOSy
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Other Study IDs: GITMO-GVCrOSy
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Chronic Graft-Versus-Host Disease
Keywords: chronic graft-versus-host disease cGVHD; Hematopoietic stem cell transplantation HSCT; NIH consensus criteria; GITMO
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cGVHD: All consecutive patients undergoing allogenic stem cell transplant for any underlying disease who develop chronic graft-versus-host disease (cGVHD)

SUMMARY:
Prospective, observational, multicentre, spontaneous, non-interventional study This study will evaluate all consecutive patients who develop chronic graft-versus-host disease, reported by the Italian GITMO centers according to a standardized Web platform for real-time, onsite data collection. The platform for data collection will be based on a software prototype developed by the Clinica di Ematologia di Ancona Transplant Center for the management of patients with chronic graft-versus-host disease. This software has been integrated with algorithms that automatically determine: severity of chronic graft-versus-host disease and overall response according to the 2015 NIH consensus criteria.

DETAILED DESCRIPTION:
Chronic Graft-versus-Host Disease represents the first cause of transplant-related mortality and reduced quality of life after transplant (HSCT). The epidemiology of Chronic Graft-versus-Host Disease is largely unknown; moreover, diagnosis of Chronic Graft-versus-Host Disease can be easily missed because its onset is often late in the post-transplant period, requires specific follow up, and general practitioners are usually not familiar with this entity. Successful treatment of Chronic Graft-versus-Host Disease represents an unmet clinical need in the field of allogeneic transplantation. Steroids are standard treatment, but up to 60% of the patients will require second-line treatment but there is no standard second-line treatment for Chronic Graft-versus-Host Disease steroid refractory. To help standardise the management Chronic Graft-versus-Host Disease, the NIH Consortium proposed consensus definitions for diagnosis, scoring and response criteria in 2006 revised in 2015 which offers a shared framework to study this rare disease. These criteria are not yet validated and thus not suitable for clinical trials.

This study is prospective, observational, multicentre, spontaneous, non-interventional study that will evaluate all consecutive patients who develop chronic graft-versus-host disease, reported by the Italian GITMO centers according to a standardized Web platform for real-time, on-site data collection. The platform for data collection will be based on a software prototype developed by the Ancona Transplant Center for the management of patients with Chronic Graft-versus-Host Disease. This software has been integrated with algorithms that automatically determine: severity of Chronic Graft-versus-Host Disease and overall response by the 2015 NIH consensus criteria. Historical controls to compare Chronic Graft-versus-Host Disease incidence, toxicities, response rate and hard outcomes will be used.

The aim of this project is to evaluate prospectively the long-term effectiveness of different therapies by the hard outcome "failure free survival" commonly considered the most reliable one. The failure free survival is the result of a number of factors that influence the treatment failure and has been shown a reliable predictor of long-term survival. Main cause of failure is the change in immunosuppressive treatment although recurrent disease, treatment toxicity and mortality from Chronic Graft-versus-Host Disease (or other infectious complications) also contribute to failure free survival. Second, we aim to evaluate the prognostic ability of the latest NIH response criteria to predict main hard survival outcomes and to assess their suitability as a tool for decision-making that ultimately leads to treatment changes. Finally, we aim to evaluate the feasibility of the use of an electronic tool for data collection in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Any age
* All patients who develop cGVHD (any grade) by the NIH criteria after allogeneic transplantation
* Written and signed informed consent

Exclusion Criteria:

* Absence of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing sllogenic stem cell transplant for any underlyng disease who develop chronic graft-versus-host disease (cGVHD)
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Failure free survival (FFS) | Measured from the start of 1st line immunosuppressive treatment for cGVHD until the date of first documented progression or date of death from any cause whichever came first, assessed up to 1 years from transplant
  To estimate the failure free survival measured from the start of 1st line immunosuppressive treatment for cGVHD, defined as the probability of survival free of any of the following events: cGVHD progression, need of a new immunosuppressive treatment, need of treatment dose escalation, relapse of the underlying hematological disease, severe (CTCAE grade 3-4) toxicity.

SECONDARY OUTCOMES:
Response rate (RR) | 3 and 6 months
  Global and organ-specific response rate (RR), evaluated 3 and 6 months after starting systemic treatment, by the 2015 NIH criteria
Incidence and grade of cGVHD | at 1 year from transplant
  Incidence and grade of cGVHD, by the 2015 NIH criteria at 1 year after Hematopoietic stem cell transplantation (HSCT)
relapse | 1 year from transplant
  Cumulative incidence of relapse of underlying haematological malignancy
non-relapse mortality | 1 year from transplant
  Cumulative incidence of non-relapse mortality (NRM), defined as any death not due to disease relapse or progression
treatment change | measured from the start of first-line and subsequent treatment lines for 1 year
  Cumulative incidence of treatment change, measured from the start of first-line and subsequent treatment lines
Successful withdrawal of immunosuppressive treatment | Measured from the start of firs-tline and subsequent treatment lines for 1 year
  Cumulative incidence of successful withdrawal of immunosuppressive treatment, measured from the start of first-line and subsequent treatment lines.
Overall Survival | measured from cGVHD diagnosis until 1 year
  Overall Survival, measured from cGVHD diagnosis.
Severe Adverse Events (SAE) and Toxicities | Measured from first treatment for cGVHD until 1 year
  Incidence of Severe Adverse Events (SAE), toxicities (by the Common Terminology Criteria for Adverse Events - CTCAE), infections during treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Attilio Olivieri, MD, Principal Investigator — AOU Ospedali Riuniti di Ancona
Locations (27):
- Italy (27):
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - Ospedale San Orsola, Bologna
  - Ospedale Regionale Generale- Divisione Ematologia, Bolzano
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - Ospedale Ferrarotto - Ematologia, Catania
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - Ospedale Gaslini, Genova
  - Osp. Card. Panico, Lecce
  - Ospedale Maggiore - Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - CTMO Fond MBBM Clinica pediatrica, Monza
  - Uoc Sit Tmo, Napoli
  - Azienda ospedaliera Universitaria di Parma, Parma
  - Ospedale G. Da Saliceto di Piacenza, Piacenza
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - Arciospedale S. M. Novella, Reggio Emilia
  - Cattedra di Ematologia - Policlinico Umberto I, Roma
  - A.O.U. Citta della Salute e della Scienza, Torino
  - Ospedale Regina Margherita, Torino
  - A.O. Santa Maria della Misericordia, Udine
  - Policlinico GB Rossi, Verona
  - Ospedale S. Bortolo-Divisione Ematologia, Vicenza